CLINICAL TRIAL: NCT00169065
Title: Clozapine vs. Olanzapine: An Effectiveness Study
Brief Title: Effectiveness of Clozapine Versus Olanzapine for Treatment-resistant Schizophrenia
Acronym: COES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Dartmouth-Hitchcock Medical Center (Other); Commonwealth Research Center, Massachusetts (Other); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, AlanGreen, Chair, Department of Psychiatry Geisel School of Medicine at Dartmouth, National Institute of Mental Health (NIMH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH049891 (NIH); R01MH049891 (NIH)
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Schizophrenia
Keywords: Clozapine; olanzapine
MeSH Terms: conditions — Schizophrenia | interventions — Clozapine; Olanzapine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clozapine (Active Comparator): Clozapine or olanzapine in treatment resistant schizophrenia
  Interventions: Drug: Clozapine
- olanzapine (Active Comparator): clozapine or olanzapine in treatment resistant schizophrenia
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Clozapine
  Arms: Clozapine
Drug: Olanzapine
  Arms: olanzapine

SUMMARY:
This study will determine the effectiveness of clozapine versus olanzapine in treating people with schizophrenia that has not improved with treatment.

DETAILED DESCRIPTION:
This is a two-year open-label, randomized trial of the comparative effectiveness of clozapine versus olanzapine in patients with treatment refractory schizophrenia. The objective is to determine whether in a naturalistic setting olanzapine is a logical treatment choice (before using the more toxic clozapine) for some treatment refractory patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60 years;
* Diagnosis of treatment refractory schizophrenia or schizoaffective disorder;
* BPRS score > 21 (0-6) scale;
* Either two 6-8 week trials of typical neuroleptics given at a dosage of 600 mg/day of CPZ or its equivalent or one 6-8 week trial of an atypical antipsychotic at a reasonable dose (i.e. risperidone 4-6 mg/day);
* The patient (or the patient's authorized legal representative) must understand the nature of the study and sign the informed consent;
* Clinically appropriate for clozapine or olanzapine

Exclusion Criteria:

* Current substance abuse;
* Suicide or homicide risk;
* Pregnancy or lactation;
* History of seizures or blood dyscrasias

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 1998-08; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Changes in quality of life.

SECONDARY OUTCOMES:
Symptom measures, neurological side effects, neuropsychological performance, patient satisfaction and burden on the family.

CONTACTS AND LOCATIONS:
Overall Officials: Alan I Green, MD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Commonwealth Research Center, Jamaica Plain, Massachusetts, United States